CLINICAL TRIAL: NCT03715517
Title: Spinal Anesthesia for Enhanced Recovery After Liver Surgery
Acronym: SAFER-L
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Alex Grunfeld, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2018:048
Record Dates: First submitted 2018-10-15; First posted 2018-10-23 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Hepatectomy; Pain, Postoperative; Liver Neoplasms
Keywords: Injections, Spinal; Analgesia, Epidural; Anesthesia, Spinal; Patient Reported Outcome Measures; Postoperative Period
MeSH Terms: conditions — Pain, Postoperative; Liver Neoplasms; Agnosia | interventions — Anesthesia, Spinal; Bupivacaine; Morphine; Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrathecal morphine (Experimental): Spinal anesthesia with intrathecal morphine
  Bolus (pre-induction): High-spinal anesthesia with 0.25 mg⋅kg-¹ hyperbaric bupivacaine 0.75% plus 3 mcg⋅kg-¹ intrathecal morphine (preservative-free)
  Postoperative analgesia: IV-PCA hydromorphone (bolus: 0.2 mg [range: 0.1-0.4 mg]; 5 min lockout; no infusion)
  Interventions: Procedure: Spinal anesthesia with intrathecal morphine; Drug: Bupivacaine 0.75% in Dextrose Inj 8.25%; Drug: Morphine
- Thoracic epidural analgesia (Active Comparator): Continuous thoracic epidural analgesia
  Bolus (pre-induction): 0.25 mg⋅kg-¹ bupivacaine 0.25% plus 1 mcg⋅kg-¹ hydromorphone (0.1 mL⋅kg-¹)
  Infusion (initial): 0.25 mg⋅kg-¹⋅h-¹ bupivacaine 0.25% plus 1 mcg⋅kg-¹⋅h-¹ hydromorphone (0.1 mL⋅kg-¹⋅h-¹)
  Infusion (range): 0.19-0. 3 mg⋅kg-¹⋅h-¹ bupivacaine 0.25% plus 0.75-1.25 mcg⋅kg-¹⋅h-¹ hydromorphone (0.075-0.125 mL⋅kg-¹⋅h-¹) (3-10 mL⋅h-¹)
  Postoperative analgesia: (1) Epidural solution, bupivacaine 0.125% with hydromorphone 10 mcg·mL-¹, infusion range as above (0.075-0.125 mL⋅kg-¹⋅h-¹) (3-10 mL⋅h-¹), continued for a maximum of 72 h postoperatively; (2) IV-PCA hydromorphone (bolus: 0.2 mg [range: 0.1-0.4 mg]; 5 min lockout; no infusion).
  Interventions: Procedure: Continuous thoracic epidural analgesia; Drug: Bupivacaine 0.25% Preservative-Free Injectable Solution; Drug: Bupicavaine 0.125% epidural solution; Drug: Hydromorphone 10 mcg/mL epidural solution

INTERVENTIONS:
Procedure: Continuous thoracic epidural analgesia — Needle/catheter: 17 Ga. × 80 mm Tuohy epidural needle (Perican®, B. Braun Medical Inc., Bethlehem, PA, USA); Arrow FlexTip Plus® 19 Ga. epidural catheter (Arrow International Inc., Reading, PA, USA)
  Level of insertion and patient positioning: T6-T8, upright sitting position for insertion of needle and catheter (to 5 cm beyond loss-of-resistance point) and for injection of test dose (3 mL 2% lidocaine with epinephrine 1:200,000); supine for injection of bolus dose
  Confirmation of correct placement: Loss of resistance to air or saline; negative aspiration of the epidural catheter; negative test dose; and ease of injection of an initial bolus dose
  Arms: Thoracic epidural analgesia
Procedure: Spinal anesthesia with intrathecal morphine — Needle/catheter: 25 Ga. × 90 mm high-flow Whitacre spinal needle (Becton-Dickinson, Franklin Lakes, NJ, USA)
  Level of insertion and patient positioning: L2-L3, lateral decubitus position during injection; immediately post-injection, patient is placed supine in <5% degree of Trendelenburg
  Confirmation of correct placement: Aspiration of cerebrospinal fluid
  Arms: Intrathecal morphine
Drug: Bupivacaine 0.75% in Dextrose Inj 8.25% — 0.25 mg⋅kg-¹ hyperbaric bupivacaine 0.75%
  Other Names: Spinal heavy bupivacaine
  Arms: Intrathecal morphine
Drug: Morphine — 3 mcg⋅kg-¹ intrathecal morphine (preservative-free)
  Other Names: Intrathecal morphine
  Arms: Intrathecal morphine
Drug: Bupivacaine 0.25% Preservative-Free Injectable Solution — 0.25 mg⋅kg-¹ bupivacaine 0.25%
  Other Names: Bupivacaine 0.25% epidural solution
  Arms: Thoracic epidural analgesia
Drug: Bupicavaine 0.125% epidural solution — Epidural solution, bupivacaine 0.125% with hydromorphone 10 mcg·mL-¹, infusion range 0.075-0.125 mL⋅kg-¹⋅h-¹
  Other Names: Bupivacaine 0.125% preservative-free injectable solution
  Arms: Thoracic epidural analgesia
Drug: Hydromorphone 10 mcg/mL epidural solution — Epidural solution, bupivacaine 0.125% with hydromorphone 10 mcg·mL-¹, infusion range 0.075-0.125 mL⋅kg-¹⋅h-¹
  Arms: Thoracic epidural analgesia

SUMMARY:
This project proposes to compare epidural versus spinal anesthesia in patients having liver resection surgery. The investigators hypothesize that spinal anesthesia will result in improved blood pressure control postoperatively and reduce the amount of intravenous fluids required after surgery. Spinal anesthesia is expected to provide the same pain control benefits as epidurals, with faster recovery of function. Spinal anesthesia may be a simple and effective way to improve and enhance the recovery in the increasing number of patients requiring liver resection.

DETAILED DESCRIPTION:
Hepatic resection surgery (hepatectomy) for primary or metastatic malignancy is a major operation involving large, painful upper abdominal incisions, as well as considerable postoperative physiological derangements.

Uncontrolled postoperative incisional pain results in significant respiratory impairment, delayed mobilization, and augmentation of the surgically-induced stress response, placing patients at increased risk of postoperative complications and chronic post-surgical pain. Acute pain management with high-dose parenteral opioids further compounds this risk. Multimodal opioid-sparing therapy, and regional anesthesia in particular, is therefore an essential component of enhanced recovery after surgery (ERAS) pathways and patient-centred care.

Regional anesthesia using neuraxial block (intraoperative spinal anesthesia or thoracic epidural anesthesia) followed by postoperative continuous thoracic epidural analgesia (CTEA; postoperative administration of epidural local anesthetic and/or opioid) is the best method for treating pain following large abdominal surgeries, including liver resection, and has been shown to improve postoperative respiratory function and decrease respiratory complications in other surgeries.

However, the effects of intraoperative neuraxial block and postoperative CTEA on fluid balance, systemic hemodynamics, and functional recovery after hepatic resection surgery remain controversial. CTEA is frequently associated with postoperative hypotension, resulting in increased perioperative intravenous (IV) fluid administration, red blood cell transfusion, and vasopressor use in liver resection patients. For major hepatectomies, CTEA may also be an independent risk factor for postoperative acute kidney injury (AKI), presumably due to impairment of renal autoregulation. Excessive IV fluid administration in the postoperative period is associated with significant weight gain, often necessitating diuretic therapy; delayed return of gastrointestinal function; increased need for packed red blood cell (pRBC) transfusion due to hemodilution; increased infective complications due to this increased pRBC transfusion rate; and increased length of hospital stay.

In addition, concerns remain about the use of CTEA following liver resection surgery due to the potentially increased risk of epidural hematoma formation in the setting of postoperative coagulopathy. This concern has resulted in unplanned delays in epidural catheter removal postoperatively, due to persistent coagulation abnormalities, prolonging hospitalization by 1-3 d in up to 15% of patients.

These concerns about the consequences of excess fluid administration and the safety of CTEA for liver resection surgery have prompted the use of alternative and/or ancillary analgesic techniques, particularly for major resections and in patients with preoperative liver dysfunction, for whom a prolonged period of postoperative coagulopathy is anticipated.

Intraoperative spinal anesthesia (SA) using local anesthetic (LA) and/or opioid (most commonly intrathecal morphine [ITM]) for neuraxial block without CTEA is frequently used as postoperative analgesia for various surgeries. Spinal anesthesia using ITM without LA has been reported in four randomized and three non-randomized studies of patients undergoing liver resections. ITM has provided superior analgesia to IV patient-controlled analgesia (IV-PCA) with opioids, and equivalent analgesia to epidural infusions. Compared with CTEA and/or IV-PCA, ITM was associated with reduced IV fluid administration; earlier mobilization, and resumption of normal dietary intake; decreased incidence of respiratory complications; and decreased hospital length of stay.

Spinal anesthesia using both LA and ITM may provide an additional benefit by providing a degree of preemptive analgesia, as well as by decreasing the stress and inflammatory response, thereby possibly decreasing the incidence of surgical stress-related complications such as postoperative delirium. High-spinal anesthesia (HSA) uses larger doses of LA to achieve a "high" block for this purpose. HSA combined with ITM has been used in cardiac surgery, and decreases the stress and inflammatory response to surgery; facilitates early extubation; improves postoperative analgesia; decreases the incidence of postoperative delirium; and decreases intensive care unit (ICU) readmissions. Neither the use of HSA (with or without ITM) for analgesia following non-cardiac surgical procedures, nor the effectiveness of SA with ITM versus CTEA following hepatic resection surgery has been investigated to date.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, Adults aged ≥ 18 years (there will be no upper age restriction);
* American Society of Anesthesiologists Physical Status classification (ASA-PS) of I to III;
* Undergoing subcostal or midline laparotomy for elective liver resection surgery under general anesthesia; if the planned procedure is a combined operation (i.e., concomitant extrahepatic surgery) , the associated procedure should not add more than one hour to the surgical time of the primary hepatic resection procedure alone;
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Provision of signed and dated informed consent form
* Body mass index (BMI) between 17 and 40 kg·m-², inclusive;
* Negative result on serum pregnancy test at Screening and negative urine pregnancy test at Baseline (for women of childbearing potential, defined as those who have not undergone a hysterectomy or been postmenopausal for at least 12 consecutive months); and not currently breastfeeding, or planning to do so within 7 d following surgery;
* Stated willingness and ability to comply with all study and/or follow-up evaluations and communicate clearly with the Investigator and staff; and
* Voluntary participation and ability to provide written informed consent prior to any study procedures.

Exclusion Criteria:

* Emergency surgery;
* Age < 18 years;
* Planned laparoscopic hepatic resection;
* Planned laparotomy incision other than (right) subcostal, midline, or extended midline;
* Patients with obvious non-resectable disease prior to signing informed consent;
* Liver transplant recipient or previous hepatic resection or living-donor hepatectomy surgery;
* Major surgery (open abdominal and/or thoracic) under general anesthesia ≤ 30 d preoperatively;
* Contraindications to neuraxial (spinal or epidural) anesthesia: (a) anticipated difficult intubation; (b) coagulation or hemostatic abnormalities within 30 d of surgery (defined as thrombocytopenia [platelet count < 100 × 10⁹ L-¹]; INR > 1.4; or activated partial thromboplastin time [aPTT] > 40 s); (c) bleeding diathesis; (d) ongoing use (≤ 7 d before surgery) or planned perioperative use of antiplatelet agents (apart from acetylsalicylic acid 81 mg) or anticoagulants (excluding deep-vein thrombosis prophylaxis); (e) recent (≤ 30 d preoperatively) systemic infection or current (≤ 48 h) fever (≥ 38.4 °C), or evidence of infection (including superficial cutaneous infection in the thoracic and/or lumbar regions); (f) history of neurologic disorder affecting the spinal cord or the hemithorax or below; or impaired bladder/bowel function; (g) acute or subacute (≤ 90 d preoperatively) intracranial hemorrhage; or (h) technical contraindications to epidural placement: (i) local skin or soft tissue infection at proposed site for thoracic epidural insertion; (ii) previous cervicothoracic, thoracic, or thoracolumbar spinal surgery; (iii) history of spinal tumor, fracture or infection; or (iv) recent (≤ 14 d preoperatively) epidural corticosteroid injection;
* Significant cardiac arrhythmias (including pacemaker-dependence) or clinically significant cardiovascular disease (New York Heart Association [NYHA] functional classification III-IV);
* Volume overload (hyperhydration), particularly in cases of pulmonary edema or acute decompensated congestive heart failure (CHF);
* Acute kidney injury (AKI) and/or chronic kidney disease (CKD) based on the 2012 Kidney Disease Improving Global Outcomes (KDIGO) AKI (excluding the oliguria criterion) and CKD guideline definitions: AKI: increase in serum creatinine (SCr) (≥ 26.5 μmol·L-¹ within 48 h or ≥ 1.5× baseline within 7 d); CKD: abnormalities of kidney structure or function, present for > 3 mo, defined as either of the following present for > 3 mo: (1) ≥ 1 marker(s) of kidney damage: (a) albuminuria (24-h albumin-creatinine ratio [ACR] ≥ 30 mg·g-¹ [≥ 3 mg·mmol-¹]), (b) urine sediment abnormalities, (c) electrolyte and other abnormalities due to tubular disorders, (d) abnormalities detected by histology, (e) structural abnormalities detected by imaging, (f) history of kidney transplantation; and/or decreased glomerular filtration rate (GFR < 60 mL-¹·min-¹·1.73 m-², estimated using the 2009 CKD-EPI creatinine equation [eGFR_creat]);
* Severe hypernatremia ([Na⁺] ≥ 155 mmol·L-¹) and/or hyperchloremia ([Cl-] ≥ 125 mmol·L-¹);
* Chronic pain; current (≤ 30 d preoperatively) and/or prior chronic (for a period of ≥ 90 d) opioid use; or history of alcohol, opiate, and/or other drug abuse or dependence;
* Use of supraphysiologic glucocorticoid (GC) doses (≥ 7.5 mg·day-¹ of prednisone or equivalent): recent (≤ 30 d), prolonged (> 2 consecutive weeks), or multiple courses totalling > 3 weeks in the preceding 6 months;
* Known allergy or sensitivity (e.g., glucose-6-phosphate dehydrogenase [G6PD] deficiency) to amide local anesthetics, opioids, or acetaminophen, or hypersensitivity to other materials to be used in the study (e.g., latex [epidural catheter adapter], epidural dressing or tape); or
* Altered mental status or educational, psychiatric, or communication (language, literacy) barriers that would impede accurate assessment of postoperative pain and/or ability to complete questionnaire instruments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2018-10-04 (Actual); Primary Completion 2031-07-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative 72-hour volume of intravenous fluids and blood products administered | Intraoperatively and during the first 72 hours postoperatively or until hospital discharge, whichever occurs earlier
  Intraoperative plus cumulative postoperative intravenous (IV) fluid volume administered, total (mL) = sum of volumes of IV crystalloid, IV colloid, and non-albumin blood products (packed red blood cells [pRBC], fresh-frozen plasma [FFP], and platelets) administered
Area under the curve over 72 hours of the summed pain intensity difference scores at rest (AUC-SPID-PAR_0-72h) | 72 hours after surgery or until hospital discharge, whichever occurs earlier
  Numerical Rating Scale (NRS) Summed Pain Intensity Difference at rest (SPID-PAR) (calculated as Area Under the Curve [AUC] using the trapezoidal rule) over 0 to 72 hours (AUC-SPID-PAR_0-72h) after surgery. Pain intensity (PI) is assessed preoperatively and at 2, 6-12, 24, 36, 48, 60, and 72 hours after surgery or until hospital discharge, whichever came first, using the 11-point Numerical Rating Scale (NRS) on a scale from 0 to 10, where 0 represents the absence of pain and 10 is the "worst possible pain". Pain intensity difference (PID_t) is calculated as the difference in pain intensity from time 0 to each time point t. SPID_t is calculated using the trapezoidal rule as the area under the curve (AUC) for Pain Intensity Difference over the time interval 0 to t hours, respectively, divided by the length of the time interval (t hours). A positive value is a decrease (improvement) of the pain.
Cumulative 72-hour opioid consumption (OC_0-72h) | Intraoperatively and during the first 72 hours postoperatively or until hospital discharge, whichever occurs earlier
  Total perioperative epidural, intravenous, and oral opioid requirements measured in oral morphine equivalents (OME, mg).

SECONDARY OUTCOMES:
Vasopressor-free days to day 30 | During index hospital admission (censored at the earliest of hospital discharge, in-hospital death, or 30 days postoperatively)
  Vasopressor-free days to 30 days after surgery will be defined as the number of days alive and not on vasopressors before 30 days. If the patient is on vasopressors at day 30 or dies prior to day 30, vasopressor-free days will be 0.
Cumulative intraoperative vasopressor and/or inotrope consumption | Intraoperatively (from anesthesia start time to anesthesia end time)
  Cumulative norepinephrine (NE)-equivalent time-weighted dose (mcg·kg-¹·min-¹ of anesthesia time) of vasopressors and/or inotropes (phenylephrine, norepinephrine, dopamine, and/or epinephrine).
Cumulative perioperative vasopressor and/or inotrope consumption | Intraoperatively and during the first 7 days after surgery or until hospital discharge, whichever occurs earlier
  Cumulative norepinephrine (NE)-equivalent time-weighted dose (mcg·kg-¹·min-¹ of vasopressor and/or inotrope infusion duration) of vasopressors and/or inotropes (phenylephrine, norepinephrine, dopamine, and/or epinephrine).
Cumulative 72-hour volume of intravenous fluids administered | Intraoperatively and during the first 72 hours postoperatively
  Intraoperative plus cumulative postoperative intravenous (IV) fluid volume administered, excluding non-albumin blood products, total (mL) = sum of volumes of IV crystalloid and IV colloid administered
Area under the curve over 72 hours of the summed pain intensity difference scores of movement-evoked pain (MEP) (AUC-SPID-MEP_0-72h) | 72 hours after surgery or until hospital discharge, whichever occurs earlier
  Numerical Rating Scale (NRS) Summed Pain Intensity Difference of movement-evoked pain (SPID-MEP) (calculated as Area Under the Curve [AUC] using the trapezoidal rule) over 0 to 72 hours after surgery (AUC-SPID-MEP_0-72h)
Cumulative incidence (proportion) of rescue analgesia (parenteral opioid) use (%) | 72 hours after surgery or until hospital discharge, whichever occurs earlier
  Rescue analgesia (parenteral opioid) use is defined as receipt of supplemental (i.e., in addition to that defined by the intervention protocols) doses of fentanyl, morphine, and/or hydromorphone via the intravenous (IV) route, either via patient-controlled analgesia (PCA) or nurse/physician administration.
Cumulative fluid balance (CFB) at 72 hours | 72 hours after surgery or until hospital discharge, whichever occurs earlier
  Cumulative fluid balance (CFB) is defined as the sum of current daily fluid balance (DFB) and the sum of DFB from all preceding days. DFB (mL) = (total daily fluid input - total daily fluid output). Daily fluid input includes: (1) resuscitation fluids (isotonic crystalloid [at a rate >1 L/6 h]; colloids [albumin, hydroxyethyl starch]); (2) blood products (packed red blood cells; frozen plasma; platelets; cryoprecipitate); (3) maintenance and replacement fluids (dextrose-containing crystalloid; isotonic crystalloid [at a rate ≤1 L/6 h]); (4) nutrition (enteral nutrition [i.e., tube feeds]; parenteral nutrition; oral fluid intake); and (5) fluid creep (volume due to concentrated electrolytes; volume used to keep venous access open; intermittent and continuous medication). Daily fluid output includes: (1) blood loss; (2) urine output; (3) dialysis ultrafiltrate (if applicable); (4) losses through drains; and (5) losses through enteric (e.g., nasogastric) tubes.
Percentage fluid overload (% FO) at 72 hours | 72 hours after surgery or until hospital discharge, whichever occurs earlier
  Percentage fluid overload (% FO) is defined as the ratio between cumulative fluid balance and the initial body weight, in percentage: % FO = [(total fluid in (L) - total fluid out (L)) / admission body weight (kg) × 100].
Volume-related weight gain (VRWG) at 72 hours | 72 hours after surgery or until hospital discharge, whichever occurs earlier
  Volume-related weight gain at time t (VRWG_t) is defined as the percentage body weight gain at time t, calculated as the difference between the baseline body weight and body weight at time t divided by baseline body weight (t = 0): VRWG_t (%) = [(body weight [kg]_t - body weight [kg]_0) / body weight [kg]_0 × 100%].
Quality of recovery, as measured by the change from baseline 15-item Quality of Recovery (QoR-15) scale score over the first 72 hours postoperatively | 72 hours after surgery or until hospital discharge, whichever occurs earlier
  Patient-reported quality of recovery (QoR), as assessed using the 15-item Quality of Recovery (QoR-15) scale, with the change from baseline in the total QoR-15 score (range 0-150) at 72 hours postoperatively defining the analysis endpoint. The QoR-15 is a 15-item patient-completed questionnaire including items measuring pain, physical comfort, psychological support, emotional state, and independence in activities of daily living over the preceding 24 hours. Items are rated on a 10-point scale, with higher subscale (item) and total scale values indicating a better outcome. The scale's validity (content, criterion, and construct), reliability (test-retest and internal consistency [inter-item and split-half coefficients]), responsiveness (minimal clinically important difference [MCID] = 8.0), acceptability, and feasibility properties have been well-established.
Time to mobilization (h) | 7 days after surgery or until hospital discharge, whichever occurs earlier
  Defined as time to first out-of-bed mobilization (sitting out of bed, standing or walking).
Time to gastrointestinal (GI) recovery (h) | 7 days after surgery or until hospital discharge, whichever occurs earlier
  Defined as the later of (1) time to solid diet tolerance (recovery of upper GI function), and (2) time to first flatus or bowel movement.
Time to removal of urinary catheter (h) | 7 days after surgery or until hospital discharge, whichever occurs earlier
Time to adequate pain control with PO medications (h) | 7 days after surgery or until hospital discharge, whichever occurs earlier
Sleep disturbance, as measured by the change from baseline Patient-Reported Outcomes Measurement Information System (PROMIS®) Short Form v1.0 - Sleep Disturbance 8a scale T-score over the first 7 days postoperatively | 7 days after surgery or until hospital discharge, whichever occurs earlier
  The Patient-Reported Outcomes Measurement Information System (PROMIS®) Short Form v1.0 - Sleep Disturbance (SD) 8a scale assesses self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. The 8-item self-report version (Short Form [SF]) of the PROMIS® SD 8a scale included in this study queries sleep disturbance symptomatology based on the past 7 days, with each item rated on a 5-point Likert scale ranging from 1 (never) to 5 (almost always). All item scores are summed to calculate a total raw score where higher scores indicate more severe sleep disturbance symptomatology. Psychometric evaluations of the 8-item PROMIS® SF SD 8a in a wide range of patient populations have provided support for its high reliability (test-retest, internal consistency) and validity (convergent, divergent, face, construct). A smaller between-group increase from baseline (preoperative) to 7-day postoperative PROMIS® SF SD 8a T-scores indicates a better outcome.
Overall Benefit of Analgesia Score (OBAS) at 72 hours | 72 hours after surgery or until hospital discharge, whichever occurs earlier
  The Overall Benefit of Analgesia Score (OBAS) is a patient-reported outcome measure of seven pain-related quality-of-life indicators: (1) pain intensity at rest (scored 0-4, 0 = minimal pain, to 4 = maximum imaginable pain); patient-reported distress with respect to five opioid-related adverse effects (each scored 0-4, 0 = not at all, to 4 = very much): (2) vomiting, (3) itching, (4) sweating, (5) freezing, and (6) dizziness; and (7) patient satisfaction with pain treatment (scored 0-4, 0 = not at all, to 4 = very much). To calculate the OBAS score, the scores for items 1-6 and 4 minus the score for item 7 are summed for a total scale score range of 0 to 28, with lower values indicating a better outcome.
Index hospitalization length of stay | During index hospital admission (censored at the earliest of hospital discharge, in-hospital death, or 30 days postoperatively)
  Duration (days) of index hospitalization from date of index operation to date of hospital discharge (censored at the earliest of hospital discharge, in-hospital death, or 30 days postoperatively).
Analgesic-related adverse events: incidence rate ratio of severe respiratory depression | During index hospital admission (censored at the earliest of hospital discharge, in-hospital death, or 30 days postoperatively)
  Severe respiratory depression is defined as respiratory rate (RR) < 8 and/or hypoxemia (Spo2 < 90%) related to excessive somnolence and/or alveolar hypoventilation.
Analgesic-related adverse events: incidence rate ratio of sedation | During index hospital admission (censored at the earliest of hospital discharge, in-hospital death, or 30 days postoperatively)
  Severe opioid-induced sedation, as defined by Pasero-McCaffery Opioid-induced Sedation Scale (POSS) score of 3 or 4. The POSS is graded on a 5-point scale (S = sleep, easy to arouse; 1 = awake and alert; 2 = slightly drowsy, easily aroused; 3 = frequently drowsy, arousable, drifts off to sleep during conversation; 4 = somnolent, minimal or no response to verbal or physical stimulation), with scores of S, 1, and 2 considered acceptable levels of sedation, and scores of 3 or 4 considered unacceptable levels of sedation.
Analgesic-related adverse events: cumulative incidence (proportion) of postoperative delirium | During index hospital admission (censored at the earliest of hospital discharge, in-hospital death, or 30 days postoperatively)
  Delirium will be evaluated via trained nursing assessments using the 3-min Confusion Assessment Method (3D-CAM). The diagnosis of delirium by 3D-CAM requires a positive response to (1) acute onset or fluctuating course; and (2) inattention; and either (3) disorganized thinking or (4) altered level of consciousness. To reduce the likelihood of fluctuations or temporal changes, all assessments were completed between 11:00 AM and 2:00 PM and for each participant, within a 2-hour time period.
Number (count) of surgical complications with Clavien-Dindo grade ≥ III | During index hospital admission (censored at the earliest of hospital discharge, in-hospital death, or 30 days postoperatively)
  Postoperative surgical complications are assessed using the Clavien-Dindo classification (none, I, II, III, IV, or V) and classified by system.
Number (count) of non-surgical complications based on the Postoperative Morbidity Survey (POMS) | Postoperative non-surgical complications are assessed using the Postoperative Morbidity Survey (POMS) based on retrospective review of medical charts and patient telephone follow-up at 30 days.
  Postoperative non-surgical complications are assessed using the Postoperative Morbidity Survey (POMS) based on retrospective review of medical charts and patient telephone follow-up at 30 days.
Comprehensive Complication Index (CCI) score Comprehensive Complication Index (CCI) score Comprehensive Complication Index (CCI) score | During index hospital admission (censored at the earliest of hospital discharge, in-hospital death, or 30 days postoperatively)
  Postoperative surgical and non-surgical complications are graded using the Comprehensive Complication Index (CCI), a continuous scale ranking the severity of any combination of postoperative complications from 0 to 100 in each patient.

OTHER OUTCOMES:
Cumulative 24-hour volume of intravenous fluids and blood products administered | Intraoperatively and during the first 24 hours postoperatively
  Intraoperative plus cumulative postoperative intravenous (IV) fluid volume administered, total (mL) = sum of volumes of IV crystalloid, IV colloid, and non-albumin blood products (packed red blood cells [pRBC], fresh-frozen plasma [FFP], and platelets) administered
Area under the curve (AUC) over 24 hours of the summed pain intensity difference (SPID) scores at rest (AUC-SPID-PAR_0-24h) | 24 hours after surgery
  Numerical Rating Scale (NRS) Summed Pain Intensity Difference at rest (SPID-PAR) (calculated as Area Under the Curve [AUC] using the trapezoidal rule) over 0 to 24 hours (AUC-SPID-PAR_0-24h) after surgery
Cumulative 24-hour (IV) opioid consumption (OC_0-24h) | Intraoperatively and during the first 24 hours postoperatively or until hospital discharge, whichever occurs earlier
  Total perioperative epidural, intravenous, and oral opioid requirements measured in oral morphine equivalents (OME, mg).
Time to first parenteral opioid dose administration (min) | 72 hours after surgery or until hospital discharge, whichever occurs earlier
  Parenteral opioid administration is defined as receipt of fentanyl, morphine, and/or hydromorphone via the intravenous (IV) route, either via patient-controlled analgesia (PCA) or nurse/physician administration.
Cumulative incidence (proportion) of patient-controlled analgesia (PCA) utilization postoperatively (%) | 7 days after surgery or until hospital discharge, whichever occurs earlier
  Patient-controlled analgesia (PCA) utilization is defined as use of PCA with intravenous opioids (morphine, fentanyl, and/or hydromorphone).
Cumulative incidence (proportion) of postoperative vasopressor and/or inotrope dependency (%) | 7 days after surgery or until hospital discharge, whichever occurs earlier
  Requirement for postoperative vasopressor and/or inotrope therapy (phenylephrine, norepinephrine, dopamine, and/or epinephrine) to maintain mean arterial pressure (MAP) ≥ 65 mm Hg and/or to treat signs and/or symptoms of systemic hypoperfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Grunfeld, MD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada